CLINICAL TRIAL: NCT02985424
Title: Polymyalgia Rheumatica and Giant Cell Arteritis - Three Challenges - Consequences of the Vasculitis Process, Osteoporosis and Malignancy: A Prospective Cohort Study Protocol
Brief Title: Polymyalgia Rheumatica and Giant Cell Arteritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Svendborg Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Amir Emamifar, Doctor of Medicine, Svendborg Hospital
Other Study IDs: S-20160098; 16/40522 (Other: Danish Data Protection Agency)
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Polymyalgia Rheumatica; Giant Cell Arteritis
MeSH Terms: conditions — Polymyalgia Rheumatica; Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: 18F-FDG PET/CT — 18F-Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography

SUMMARY:
The purpose of this study is to delineate the association of the 18F-Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography (18F-FDG PET/CT) detected vasculitis pattern of the large vessels (PET positivity) and the clinical picture of Polymyalgia Rheumatica (PMR)/Giant Cell Arteritis (GCA) .

DETAILED DESCRIPTION:
Introduction:

Polymyalgia Rheumatica (PMR) and Giant Cell Arteritis (GCA) are common inflammatory conditions. The diagnosis of PMR/GCA poses many challenges since there are no specific diagnostic tests. Recent literature emphasizes the ability of 18F-Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography (18F-FDG PET/CT) to assess global disease activity and/or inflammation burden. 18F-FDG PET/CT may lead to make diagnosis at an earlier stage than conventional imaging and assess response to therapy. With respect to the management of PMR/GCA, there are three significant areas of concern as follows: Vasculitis process/vascular stiffness, malignancy and osteoporosis.

Methods and Analysis:

Patients: All patients with the suspicion of PMR/GCR will be offered to participate in the study. The current protocol consists of 4 separate studies including: I) The association of clinical picture of PMR/GCA with PET detected vasculitis II) Evaluating validity of 18F-FDG PET/CT scan for diagnosis of PMR/GCA compared to temporal artery biopsy III) Incidence of new diagnosed malignancies in patients with PMR/GCA, or PMR like syndrome with the aim of PET/CT scan and Chest X ray/Abdominal ultrasound IV) Impact of disease process as well as steroid treatment on bone mineral density, body composition and vasculitis/vascular stiffness in PMR/GCA patients.

ELIGIBILITY:
Inclusion Criteria:

* At least five (A-E) components of the PMR diagnostic criteria, including:

  * A. Age ≥50 years,
  * B. Bilateral shoulder or hip pain,
  * C. Morning stiffness lasting >45 min,
  * D. Elevated erythrocyte sedimentation rate (ESR),
  * E. Elevated C-reactive protein (CRP),
  * F. Disease duration >2weeks, should be met to suspect PMR.
* For GCA following criteria's must be seen: Age > 50 years, ESR/CRP > 50, as well as at least two symptoms related to vasculitis (scalp tenderness, vision disturbances, headache (new or changed), jaw claudication, tenderness of the temporal arteria) if patients do not simultaneously have PMR. If the patient is suspected for PMR, one cranial symptom is enough to suspect GCA.

Exclusion Criteria:

* Dementia
* Inability to communicate in Danish
* Infections or malignancy when prednisolone is permanently unsuitable
* Contraindication to imaging studies (allergy to contrast materials, reduced kidney function, pregnancy and Blood Sugar (BS) >8 mmol/l after 6 hours fasting)
* Initiation of steroid treatment before the PET scan
* Inability to provide informed consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All new patients with clinical suspicion of PMR/GCA.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Cumulated prednisolone dose within the first year after treatment initiation in patients with and without vasculitis in the large vessels | One year

SECONDARY OUTCOMES:
Patient reported global visual analogue scale (VAS) in patients with vasculitis in the large vessels (positive PET) | One year
  Patient global assessment of disease severity as measured on a visual analogue scale (VAS) that ranges from 0 to 100, in patients with vasculitis in the large vessels detected by PET scan
Physician reported visual analogue scale (VAS) in patients with vasculitis in the large vessels (positive PET) | One year
  Physician assessment of disease severity as measured on a visual analogue scale (VAS) that ranges from 0 to 100 in patients with vasculitis in the large vessels detected by PET scan.
Patient reported pain in patients with vasculitis in the large vessels (positive PET) | One year
  Patient assessment of pain intensity as measured on a visual analogue scale (VAS) that ranges from 0 to 100, in patients with vasculitis in the large vessels detected by PET scan
Morning stiffness (minute) in patients with vasculitis in the large vessels (positive PET) | One year
Biochemistry results in patients with vasculitis in the large vessels (positive PET) | One year
  ESR, CRP and fibrinogen
Number of relapses in patients with vasculitis in the large vessels (positive PET) | One year
Proportion of PET positivity (vasculitis in the large vessels as well as findings compatible with PMR) in patients with temporal artery biopsy positive. | One year
Proportion of PET negativity (no signs of vasculitis in the large vessels) in patients with temporal artery biopsy negative. | One year
Incidence of malignancies in the included patients detected by the aim of 18F-FDG PET/CT scan. | One year
Incidence of malignancies in the included patients detected by the aim of Chest X Ray plus abdominal Ultrasound. | One year
Impact of disease process and steroid treatment on Aortic Pulse Wave Velocity (PWV) | One year
Impact of disease process and steroid treatment on upper limb PWV | One year
Impact of disease process and steroid treatment on Aortic augmentation index | One year
Impact of disease process and steroid treatment on Body Mass Index | One year
Impact of disease process and steroid treatment on T score | One year
Impact of disease process and steroid treatment on Z score | One year
Impact of disease process and steroid treatment on Lean Body Mass | One year
Impact of disease process and steroid treatment on Fat Mass | One year
Impact of disease process and steroid treatment on Bone Mineral Density | One year
Impact of disease process and steroid treatment on Bone Mineral Content | One year
Impact of disease process and steroid treatment on Fat Free Mass | One year
Impact of disease process and steroid treatment on Fat Free Mass Index | One year
Impact of disease process and steroid treatment on Fat Mass Index | One year

CONTACTS AND LOCATIONS:
Overall Officials: Inger Marie Jensen Hansen, Phd, DMSci, Study Chair — Department of Rheumatology, Odense University Hospital, Svendborg Hospital, Svendborg, Denmark.
Locations (1):
- Department of Rheumatology, Odense University Hospital, Svendborg Hospital, Svendborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Emamifar A, Hess S, Ellingsen T, Gerke O, Ahangarani Farahani Z, Syrak Hansen P, Jensen Hansen IM, Thye-Ronn P. Clinical presentation and treatment response in patients with polymyalgia rheumatica and giant cell arteritis during a 40-week follow-up. Rheumatol Adv Pract. 2021 Nov 24;5(3):rkab091. doi: 10.1093/rap/rkab091. eCollection 2021. PMID 34909566